CLINICAL TRIAL: NCT05316805
Title: China Type II Inflammatory Skin Disease Clinical Research and Standardized Diagnosis and Treatment Project: a National Multicenter Prospective Cohort Study
Brief Title: China Type II Inflammatory Skin Disease Clinical Research and Standardized Diagnosis and Treatment Project
Acronym: CORNERSTONE
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PKU202108
Record Dates: First submitted 2022-03-18; First posted 2022-04-07 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Atopic Dermatitis Eczema; Prurigo Nodularis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In order to further improve the diagnosis and treatment level of type 2 inflammatory skin diseases, the National Clinical Center for Skin and Immune Diseases established a standardized diagnosis and treatment center for type 2 inflammatory skin diseases to systematically and effectively understand the current treatment status of patients with type 2 inflammatory skin diseases, as well as the efficacy and safety of various treatment methods during practices, so as to further improve the diagnosis and treatment level of type 2 inflammatory skin diseases and help patients with type 2 inflammatory skin diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients from the medical units that has passed the data review of the National Clinical Center for Skin and Immune Diseases (see the study sites for data collection for details);
2. patients diagnosed with type 2 inflammatory skin diseases (dermatitis/eczema, urticaria, pemphigoid, prurigo nodularis).

Exclusion Criteria:

1. patients who fail to provide informed consent form;
2. patients who cannot complete the questionnaire independently or under the guidance of investigators

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Type 2 skin disease. Estimated number of patients: 100,000 (No age limit)
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2021-08-31 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Demographics | baseline
  Age, sex, ethnicity, body weight and height
Age at Type 2 skin disease onset | baseline
  Age of study patients at time of Type 2 skin disease onset
Type of current Type 2 skin disease therapy | Baseline
  Type of therapy administered to treat Type 2 skin disease (e.g., systemic, topical, other)
Presence of Type 2 skin disease and selected comorbid conditions | Baseline to Month 120
  Percentage of patients with Type 2 skin disease and selected comorbidities (e.g., asthma and allergic rhinitis) at baseline and during study

SECONDARY OUTCOMES:
Percentage of patients using specific Type 2 skin disease therapies and initiating new therapies | Baseline to Month 120
  Percentage of patients using specific Type 2 skin disease therapies and initiating new therapies
Eczema Area and Severity Index (EASI) | Baseline to Month 120
  EASI score as assessed by physician
Body Surface Area (BSA) percentage affected by Type 2 skin disease | Baseline to Month 120
  BSA score as assessed by physician
Patient Oriented Eczema Measure (POEM) questionnaire | Baseline to Month 120
  POEM score as reported by the participant's caregiver
Dermatology Life Quality Index | Baseline to Month 120
  DLQI score as reported by the patients or caregivers
Bullous Pemphigoid Disease Area Index(BPDAI) | Baseline to Month 120
  BPDAI score as assessed by physician
Autoimmune Bullous Skin Disorder Intensity Score (ABSIS) | Baseline to Month 120
  ABSIS score as assessed by physician
Chronic Urticaria Quality of Life questionnaire (CU-Q2oL) | Baseline to Month 120
  CU-Q2oL score as assessed by patients or caregivers
Urticaria Activity Score 7a （UAS7a） | Baseline to Month 120
  UAS7a score as assessed by physician
Urticaria Control test (UCT) | Baseline to Month 120
  UCT score as assessed by patients or caregivers

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhao J, Zhang Z, Chen H, Dou X, Zhao Z, Liu L, Wang Y, Li H. Associations of demographics, aggravating factors, comorbidities, and treatments with atopic dermatitis severity in China: A national cross-sectional study. Chin Med J (Engl). 2024 Mar 3;138(5):553-561. doi: 10.1097/CM9.0000000000003042. Epub 2024 Mar 3. PMID 38431766